CLINICAL TRIAL: NCT02209194
Title: PLIANT - A Post-market Registry in Patients With Iliac Aneurysm Undergoing Endovascular Stenting With a New Generation of Low Profile E-liac Stent Graft System
Brief Title: Post-market Registry in Patients With Iliac Aneurysm Undergoing Endovascular Stenting With the E-liac Stent Graft System
Status: Completed | Type: Observational
Sponsor: JOTEC GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: PLIANT
Record Dates: First submitted 2014-07-30; First posted 2014-08-05 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Iliac Aneurysm
Keywords: aneurysms; vascular disease; E-liac Stent Graft; E-liac Stent Graft System; iliac aneurysm; branched stent graft; self expanding stent graft
MeSH Terms: conditions — Iliac Aneurysm; Aneurysm; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aortoiliac Aneurysms Iliac Aneurysms: Endovascular repair of aortoiliac or iliac aneurysms
  Interventions: Device: E-liac Stent Graft System

INTERVENTIONS:
Device: E-liac Stent Graft System — Implantation of the E-liac Stent Graft System in combination with a peripheral covered stent and in case of aortoiliac aneurysm in combination with a AAA Stent Graft

SUMMARY:
The purpose of the study is to evaluate the clinical and technical success as well as safety and feasibility of the E-liac Stent Graft System used in endovascular treatment of uni- or bilateral aortoiliac or iliac aneurysm. Main study target is the exclusion of aneurysm with primary patency of the arteria iliaca interna and the arteria iliaca externa on iliac implantation side.

ELIGIBILITY:
Inclusion Criteria:

* Patients must comply with the indications for use
* Unilateral or bilateral common iliac aneurysm diameter equal or greater 25mm
* Unsuitable distal sealing site within the common iliac artery for traditional EVAR

Exclusion Criteria:

* Patients with a stenotic internal iliac ostium of < 4mm in diameter
* Patients with severe internal iliac atherosclerosis
* Patients that do not have a suitable landing area in the main stem of the IIA
* Patients with pseudoaneurysms
* Patients with symptomatic and ruptured iliac aneurysms
* Patients with one of the contraindications as indicated in the instructions for use
* Patients pretreated with a bifurcated vascular graft
* Patient with thrombocytopenia
* Patient with creatinine >2.4 mg/dl immediately before the intervention
* Patient with malignancy needing chemotherapy or radiation
* Patients who are enrolled in another clinical study
* Patients with life expectancy of less than 36 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with uni- or bilateral aortoiliac or common iliac aneurysm
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2014-06; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Primary patency | within 30 days
  Primary patency of the arteria iliaca interna and the arteria iliaca externa on E-liac implantation side
Primary Patency | 12 months
Primary patency | 36 months
Endoleak Type I or III | within 30 days
Endoleak Type I or III | 12 months
Endoleak Type I or III | 36 months

SECONDARY OUTCOMES:
Change in aneurysm size | within 30 days (baseline) and 36 months
Stent graft migration | within 30 days (baseline) and 36 months
Stent graft dislodgement | 36 months
Stent graft kinking | 36 months
Distal embolization | 36 months
Rate of death | 36 months
Rate of complications | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan Brunkwall, Professor, Principal Investigator — Cologne University Hospital
Locations (12):
- Austria (2):
  - Herzzentrum Hietzing, Vienna
  - Wilhelminenspital, Vienna
- Germany (7):
  - German Heart Center, Berlin
  - Klinikum Chemnitz, Chemnitz
  - Cologne University Hospital, Cologne
  - Uniklinikum Düsseldorf, Düsseldorf
  - UKSH Campus Kiel, Kiel
  - Krankenhaus Leonberg, Leonberg
  - Marienhospital, Osnabrück
- Instytut Hematologii i Transfuzjologii, Warsaw, Poland
- Spain (2):
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Clínico Universitario de Valladolid, Valladolid

REFERENCES:
- [Background] Brunkwall JS, Vaquero-Puerta C, Heckenkamp J, Egana Barrenechea JM, Szopinski P, Mertikian G, Seifert S, Rumenapf G, Buz S, Assadian A, Majd P, Mylonas S, Calavia AR, Theis T, de Blas Bravo M, Pleban E, Schupp J, Esche M, Kocaer C, Hirsch K, Oberhuber A, Schafer JP. Prospective Study of the Iliac Branch Device E-liac in Patients with Common Iliac Artery Aneurysms: 12 Month Results. Eur J Vasc Endovasc Surg. 2019 Dec;58(6):831-838. doi: 10.1016/j.ejvs.2019.06.020. Epub 2019 Oct 12. PMID 31615695
- [Background] Brunkwall J, Vaquero Puerta C, Heckenkamp J, Egana Barrenechea JM, Szopinski P, Mertikian G, Seifert S, Rumenapf G, Buz S, Assadian A, Majd P, Mylonas S, Revilla Calavia A, Theis T, de Blas Bravo M, Pleban E, Schupp J, Esche M, Kocaer C, Hirsch K, Oberhuber A, Schafer JP. Prospective study of the E-liac Stent Graft System in patients with common iliac artery aneurysms: 30-Day results. Vascular. 2018 Dec;26(6):647-656. doi: 10.1177/1708538118789510. Epub 2018 Jul 23. PMID 30037302
- [Background] Anton S, Wiedner M, Stahlberg E, Jacob F, Barkhausen J, Goltz JP. Initial Experience with the E-liac(R) Iliac Branch Device for the Endovascular Aortic Repair of Aorto-iliac Aneurysm. Cardiovasc Intervent Radiol. 2018 May;41(5):683-691. doi: 10.1007/s00270-017-1868-x. Epub 2018 Jan 3. PMID 29299625
- [Background] Mylonas SN, Rumenapf G, Schelzig H, Heckenkamp J, Youssef M, Schafer JP, Ahmad W, Brunkwall JS; E-liac Collaborative Group. A multicenter 12-month experience with a new iliac side-branched device for revascularization of hypogastric arteries. J Vasc Surg. 2016 Dec;64(6):1652-1659.e1. doi: 10.1016/j.jvs.2016.04.065. Epub 2016 Aug 1. PMID 27492764